CLINICAL TRIAL: NCT04399785
Title: Phase II Study for Combination of Camrelizumab and Stereotacic Radiotherapy in the First-line Treatment for Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Phase II Study for Combination of Camrelizumab and SBRT in the First-line Treatment for R/M HNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xingchen Peng (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Xingchen Peng, Associate professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CART0326
Record Dates: First submitted 2020-05-16; First posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Anti-PD-1 Inhibitor; Stereotacic Radiotherapy; Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Combination of camrelizumab and stereotacic radiotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Other: Camrelizumab and SBRT

INTERVENTIONS:
Other: Camrelizumab and SBRT — Camrelizumab: 200mg every 3 weeks; SBRT

SUMMARY:
This study is a prospective, single-center, open-label, phase II clinical study for patients with recurrent or metastatics quamous cell carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the head and neck;
2. Patients with untreated recurrent or metastatic disease;
3. Combined positive Score>=1;
4. Aged >=18 years;
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;
6. At least one measurable lesion, according to RECIST 1.1;
7. Major organ functions within 28 days prior to treatment meet the following criteria(14 days without transfusion):

   1. HB>=80g/L, ANC>=1.5x10^9/L, PLT >=80x10^9/L;
   2. TBIL<=1.5 ULN, ALT and AST <=2.5 ULN, if there exists hepatic metastases, ALT and AST <=5 ULN, Cr <=1.5 ULN or CCr >=60ml/min;
   3. INR or PT <= 1.5 ULN, APTT <=1.5 ULN (if the patient is receiving anticoagulant therapy, PT and APTT should be within the expected treatment range);
   4. BNP <=ULN;
   5. T3 <=ULN and T4 <=ULN after treatment;
8. Appropriate contraception should be used from the start of treatment to 120 days after the end of treatment; For female subjects with reproductive potential: a negative serum pregnancy test;
9. Have signed consent form.

Exclusion Criteria:

1. Have other malignant tumors in the past 5 years, except for cured in cured basal cell carcinoma, situ cervical carcinoma and thyroid papillary carcinoma ;
2. Known allergic reactions to the components of PD-1 monoclonal antibody;
3. Central nervous system metastasis with symptoms;
4. Treatment with a strong CYP3A4 inhibitor within 1 week or a strong inducer of CYP3A4 within 2 weeks.
5. Congestive heart failure of New York Heart Association (NYHA) Class III or IV;
6. Ischemic cardiovascular events occurred within 1 year prior to the start of treatment;
7. ECG QT interval >500ms;
8. Patients are receiving immunosuppressive therapy;
9. Treatment with an immunotherapy, including anti-PD-1, anti-PD-L1 and anti-CTLA-4;
10. Treatment with an investigational agent within 4 weeks;
11. Treatment with oral or parenteral corticosteroids (>10mg per day) within 2 weeks or a requirement for chronic systemic immunosuppressive therapy;
12. Treatment with anti-tumor vaccine or live vaccines within 4 weeks
13. Surgery or severe trauma within 4 weeks;
14. Active infection;
15. Active autoimmune disease;
16. History of immunodeficiency, including HIV antibody positive, primary immunodeficiency, or the allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
17. History of noninfectious pneumonia;
18. Active tuberculosis within 1 year, or had a history of active tuberculosis infection one year ago but did not receive standard treatment;
19. Active hepatitis, including HBV DNA ≥ 2000IU/ml or 10 ⁴ copies / ml or HCV antibody and HCV-RNA positive;
20. History of alcoholism and drug abuse;
21. Patients with symptoms of gastrointestinal bleeding or risk of bleeding;
22. Patients are pregnant or breast-feeding;
23. Any other condition or circumstance that could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
ORR | up to approximately 2 years
  Objective Response Rate

SECONDARY OUTCOMES:
PFS | up to approximately 2 years
  Progression-Free-Survival
OS | up to approximately 2 years
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up
DOR | up to approximately 2 years
  Disease Control Rate
AE | from the first drug administration to within 30 days for the last therapy
  Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Xingchen Peng, Chengdu, Sichuan, China